CLINICAL TRIAL: NCT01755572
Title: Hormonal Regulation of Systolic Blood Pressure in Response to the GLP-1 (Glucagon-Like Peptide-1) Receptor Agonist, Liraglutide.
Brief Title: Blood Pressure Outcomes With Liraglutide Therapy
Acronym: BOLT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: MSH-12-0020-A
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes; Systolic Hypertension
Keywords: Type 2 Diabetes; Hypertension; Liraglutide; GLP-1
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Isolated Systolic Hypertension; Hypertension | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liraglutide (Experimental): Liraglutide 0.6mg for 7 days, liraglutide 1.2mg for 7 days, liraglutide 1.8mg for 7 days
  Interventions: Drug: Liraglutide; Drug: Placebo
- Placebo (Placebo Comparator): Placebo 0.6mg sc for 3 weeks, Placebo 1.2mg sc for 3 weeks, Placebo 1.8mg for 3 weeks.
  Interventions: Drug: Liraglutide; Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide — Single cross-over study, 1 arm starting with liraglutide for 3 weeks crossed-over to placebo for 3 weeks, and 1 arm starting with placebo with cross-over to liraglutide for 3 weeks.
  Other Names: Victoza
Drug: Placebo — Single cross-over study, 1 arm starting with liraglutide for 3 weeks crossed-over to placebo for 3 weeks, and 1 arm starting with placebo with cross-over to liraglutide for 3 weeks.

SUMMARY:
Purpose:

The purpose of this study is to further study the mechanism by which liraglutide, a relatively new anti-hyperglycemic medication, might lower blood pressure in patients with Type 2 diabetes and high blood pressure.

DETAILED DESCRIPTION:
Background: Type 2 diabetes is a worldwide health problem. As the reduction in blood pressure has been coupled to improvements in overall cardiovascular outcomes, the control of hypertension has become an important modifiable risk factor in the overall care of the patient with Type 2 Diabetes, in addition to glycemic control. Recently, several large-scale clinical trials evaluating the glucose-lowering effects of the anti-hyperglycemic agent, liraglutide (a glucagon-like peptide-1 receptor agonist), have demonstrated a modest yet persistent anti-hypertensive effect in patients with Type 2 diabetes.

Study Objectives: Accordingly, the goal of this small study is to understand whether the blood pressure lowering effect of liraglutide is coupled to the release of vasoactive mediators which may stimulate natriuresis and/or diuresis and lower systolic blood pressure.

Study Design: Randomized, double-masked, cross-over study with treatment of liraglutide or placebo for 3 weeks, with an intervening washout period for 3 weeks, and cross-over to identical treatment with placebo or liraglutide for 3 weeks.

Study Patients: 20 patients with Type 2 Diabetes and Systolic Hypertension

Endpoints: Change in vasoactive hormones, 24-hour ambulatory blood pressure, urinary sodium excretion patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between the ages of 30-70.
2. Patients with Type 2 Diabetes [diagnosed by their physician] with a serum HbA1c ≥ 6.5% and ≤ 10%.
3. Patients currently prescribed 0-2 oral hypoglycemic agents by their physician.
4. Patients with systolic blood pressure ≥ 130 mmHg and ≤ 180 mmHg measured by an automated oscillometric blood pressure device [BPTru® or DinaMAP®].

Exclusion Criteria:

1. Individuals with Type 1 Diabetes, [or secondary forms of diabetes including gestational diabetes, transplant-associated, glucocorticoid-associated, latent-onset diabetes of the adult, or known monogenic forms of diabetes].
2. Elevated LVEDP (left ventricular end-diastolic pressure) including congestive heart failure, cardiomyopathy, atrial fibrillation, any valvular heart disease (rated by echocardiography and/or clinically by a cardiologist as moderate or severe in nature), and or elevated RVEDP (right ventricular end-diastolic pressure) including pulmonary hypertension.
3. Moderate renal failure or dysfunction as indicated by a serum creatinine >150 μmol/l, and/or an estimated GFR (Glomerular Filtration Rate) less than 59 ml/min per 1.73m2.
4. Individuals with secondary forms of hypertension including primary hyperaldosteronism, renal artery stenosis, obstructive sleep apnea, pheochromocytoma, hyperthyroidism, acromegaly, exogenous systemic glucocorticoid use, hypercortisolism.
5. Current pregnancy, or recent pregnancy within the last 3 months, or current breast-feeding. Female patients of child bearing potential [premenopausal, or not surgically sterile] who are unwillingly to have a baseline serum pregnancy test, and/or who are unwillingly to use active contraception throughout the duration of the study.
6. Use within the last 3 months of any DPP-IV (Dipeptidyl Peptidase) inhibitor, GLP-1 receptor agonist [liraglutide, exenatide (ExBID, or Ex QW)], or insulin [bolus, pre-mixed, or prandial].
7. Liver failure, including liver cirrhosis or non-alcoholic fatty liver disease.
8. Dependence upon alcohol, >14 servings per week if male, >9 servings per week if female.
9. Prior history of any clinical presentation consistent with pancreatitis [acute or chronic], or a history of medullary thyroid cancer, c-cell hyperplasia or history of multiple endocrine neoplasia syndromes which predisposes to medullary thyroid cancer [Multiple Endocrine Neoplasia Type 2].
10. Individuals with severe systolic hypertension, SBP (systolic blood pressure) ≥ 181 mmHg measured by an automated oscillometric blood pressure device [BPTru® or DinaMAP®].
11. Individuals with severe diastolic hypertension, DBP (diastolic blood pressure) ≥ 100 mmHg measured by an automated oscillometric blood pressure device [BPTru® or DinaMAP®].
12. Individuals currently prescribed an insulin secretagogue [sulphonylurea] unwillingly to decrease their dose by 50% prior to the start of, and for the duration of the study.
13. Individuals with resting tachycardia of >100 bpm or individuals who have a prior history of known conduction abnormalities associated with tachycardia including atrial fibrillation, atrial flutter, prolongation of PR interval, or ventricular tachycardias.
14. Current involvement, or any recent involvement [within 3 months] in any other clinical trial involving an investigational product.
15. Unwillingness to perform daily sc injection with study drug therapy for duration of 21 days throughout 2 treatment phases.
16. Individuals who are currently taking or who have taken diuretic therapy in the past 3 months.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in plasma ANP level at 1 Day | Change from Baseline compared in plasma ANP following 1 dose of liraglutide (0.6 mg) compared to crossover treatment with placebo at the 2-hour timepoint
  +16.72 pg/mL, P = 0.24, 95% CI [-12.1, +45.5] at 2 hours
Change in plasma ANP level at 21 Days | Change from Baseline in plasma ANP following 21 days of liraglutide (titrated to 1.8 mg) compared to crossover treatment with placebo at the 2-hour timepoint
  -17.42 pg/mL, 95% CI [-36.0, +1.21] at 2 hours

SECONDARY OUTCOMES:
Change in mean 24-Hr urinary sodium excretion rate following 21 days of liraglutide (titrated 1.8mg) compared to crossover with placebo (baseline-subtracted) | 21 days
  median change +14.18 mmol/L liraglutide vs. placebo (statistically significant, Wilcoxon rank sum)
Change in mean Nighttime urinary sodium excretion rate following 21 days of liraglutide (titrated 1.8mg) compared to crossover with placebo (baseline-subtracted) | 21 days
  median change +4.24 mmol/L nighttime, liraglutide vs. placebo (statistically significant, Wilcoxon Rank Sum)
Change in mean 24-Hr systolic BP, liraglutide compared to crossover with placebo (baseline-subtracted) | 21 days
  +2.33 ± 1.67, p=0.18;Treatment difference liraglutide (1.8 mg) vs. placebo LSMD (±SE), p value
Change in mean 24-hr diastolic BP, liraglutide compared to crossover with placebo (baseline-subtracted) | 21 days
  +3.78 ± 1.34, p=0.01;Treatment difference liraglutide (1.8 mg) vs. placebo LSMD (±SE), p value
Change in mean 24-hr HR, liraglutide compared to crossover with placebo (baseline-subtracted) | 21 days
  +5.21 ± 2.42, p=0.05; Treatment difference liraglutide (1.8 mg) vs. placebo LSMD (±SE), p value
Office-measured systolic BP; Treatment difference for liraglutide compared to crossover with placebo | 21 days
  -2.35 mmHg (3.49), p=0.51;Treatment difference liraglutide (1.8 mg) vs. placebo LSMD (±SE), p value
Office-measured diastolic BP;Treatment difference for liraglutide compared to crossover with placebo | 21 days
  +3.6 mmHg (2.33), p=0.14;Treatment difference liraglutide (1.8 mg) vs. placebo LSMD (±SE), p value
Office-measured heart rate;Treatment difference for liraglutide compared to crossover with placebo | 21 days
  +9.25 (3.51), p=0.02;Treatment difference liraglutide (1.8 mg) vs. placebo LSMD (±SE), p value

OTHER OUTCOMES:
Change in HbA1c% | 21 days
  -0.7%, p=0.005; least squares mean difference, liraglutide compared placebo
Change in Fasting Blood Glucose | 21 days
  -3.4 mmol/L, p=0.0004; least squares mean difference, liraglutide compared to crossover with placebo, p-value
Change in Total Cholesterol | 21 days
  -0.63 mmol/L, p=0.002; least squares mean difference, liraglutide compared to crossover with placebo, p-value
Change in LDL Cholesterol | 21 days
  -0.37 mmol/L, p=0.04; least squares mean difference, liraglutide compared to crossover with placebo, p-value
Change in eGFR (estimated Glomerular Filtration Rate) | 21 days
  -5.76 ml/min/1.73m2 (2.60), p=0.04; least squares mean difference, liraglutide compared to crossover with placebo, (SE), p-value
Change in Body Weight | 21 days
  +1.35 Kg (0.46), p=0.009; least squares mean difference (SE), p-value, liraglutide compared to crossover with placebo
Change in BMI (Body Mass Index) | 21 days
  -0.42 Kg/cm2 (0.18), p=0.03; least squares mean difference (SE), p-value, liraglutide compared to crossover with placebo
Change in Plasma Angiotensin II | 21 days
  -0.97 pmol/L (0.86), p=0.28; least squares mean difference (SE), p-value, liraglutide compared to placebo
Change in Plasma CRP | 21 days
  0.09 mg/L (0.80), p=0.91; least squares mean difference (SE), p-value, liarglutide compared to placebo
Change in Triglycerides | 21 days
  -0.2 mmol/L (0.18), p=0.28;least squares mean difference (SE), p-value, liarglutide compared to placebo
Change in HDL | 21 days
  +0.083 mmol/L (0.03), p=0.02;least squares mean difference (SE), p-value, liarglutide compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Daniel J. Drucker, MD, Principal Investigator — Samuel Lunenfeld Research Institute; Dr. Julie A. Lovshin, MD, PhD, Study Director — Samuel Lunenfeld Research Institute; Dr. Bernard Zinman, MD, Study Director — Leadership Sinai Centre for Diabetes; Dr. Alexander A. Logan, MD, Study Director — Samuel Lunenfeld Research Institute
Locations (1):
- Leadership Sinai Centre for Diabetes, Mount Sinai Hospital, Canada, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lovshin JA, Barnie A, DeAlmeida A, Logan A, Zinman B, Drucker DJ. Liraglutide promotes natriuresis but does not increase circulating levels of atrial natriuretic peptide in hypertensive subjects with type 2 diabetes. Diabetes Care. 2015 Jan;38(1):132-9. doi: 10.2337/dc14-1958. Epub 2014 Nov 20. PMID 25414155